CLINICAL TRIAL: NCT05308303
Title: Using Artificial Intelligence to Improve Data From Danish Cardiac Arrest Registry
Brief Title: AI to Improve Data From Danish Cardiac Arrest Registry
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Prehospital Center, Region Zealand (Other)
Responsible Party: Principal Investigator, Signe Amalie Wolthers, MD, principal investigator, Prehospital Center, Region Zealand
Other Study IDs: AI_CA_2022
Record Dates: First submitted 2022-02-24; First posted 2022-04-04 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Trauma; Drug Overdose; Electrocution; Asphyxia; Airway Obstruction
Keywords: Out-of-Hospital Cardiac Arrest of non-cardiac origin; traumatic Cardiac Arrest; Drug Overdose; Electrocution; Asphyxia; Cardiopulmonary Resuscitation; Emergency Medical Service
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Wounds and Injuries; Drug Overdose; Asphyxia; Airway Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- All cause OHCA
- OHCA of non-cardiac origin

SUMMARY:
Out-of-hospital cardiac arrest is a leading cause of death worldwide and patient outcome vary substantially throughout regions suggesting further evaluation and potential for improvement.When focussing on subgroups of OHCA, data in certain areas remains scarce and the need of revised guidelines is evident. Furthermore, enhanced knowledge on these varieties of OHCA's apply to substantial number of patients, also among vulnerable populations. The Danish Emergency Medical System introduced a nationwide registry of electronic medical reports in 2016. This report system allows electronic searches and thereby the opportunity to identify subgroups of OHCA's. Thus, this novel reporting enables the evaluation of new characteristics of cardiac arrests of non-cardiac origin, in cases where an automated external defibrillator (AED) is retrieved but did not recommend defibrillation and finally in OHCA related to foreign body obstruction. With the advantages of artificial intelligence, this project will enhance and strengthen data from the Danish Cardiac Arrest Registry. It may substitute the manual validation of the around 9000 cases per year in Denmark. Further, it proposes improvement of quality and development of observational health research.

DETAILED DESCRIPTION:
OHCA of non-cardiac origin is a heterogenous subgroup within a range of causes including trauma, electrocution, asphyxia (external), drowning and drug overdose. This classification of presumed etiology accounts for up to 40% of all OHCA's, but varying rates have been reported also advocating for standardised reporting and coherence to the Utstein reporting template.Compared to OHCA's with presumed cardiac etiology, the group of non-cardiac etiology has been associated with a worse prognosis.(7,9) Increased effort has been put into improvement in both prehospital and in-hospital treatment during the last two decades, but morbidity and mortality remains high with reported survival rates of around 10%. The Utstein recommendations have, since the establishment in 1991 undergone revisions in 2004 and 2015.Through the progress and revisions of the Utstein reporting template, registries have emerged worldwide; systematic reporting is, however still lacking. Besides that, most data within the field of OHCA is on cases with presumed cardiac cause.

With aid of machine learning, the hypothesis is that advances text searches may lead to improvement of quality of data from the Danish registry of OHCA. With this improvement this project might contribute to the handling and strategies concerning defined subgroups within OHCA.

Furthermore, we speculate that this novel data from the EMS medical reports provide new and central data reversible on causes, which presumably are linked to enhanced survival of OHCA of non-cardiac origin. Thus, this study aims to:

* Investigate descriptives of traumatic out-of-hospital cardiac arrest, drug overdose, electrocution and external asphyxia leading to cardiac arrest
* Assess outcomes of cardiac arrests of non-cardiac origin
* Evaluate inter- and intrasystem comparisons

Data on OHCA's with attempted resuscitation in Denmark have been collected in the electronic based Danish Medical Service reporting system since 2016. The registry covers detailed data including the EMS report. The data consists of executive entries and advanced text searches of prehospital charts in conjunction, augmenting the identification and collecting all OHCA's in Denmark. All cases have been through an elaborate validation process of which all identified events were read through manually. This was conducted by an external verification team to corroborate high quality of data throughout the approximately 5400 cases of OHCA in Denmark annually. Within this practice of verification, supplementary sources of data have been linked to each individual case of OHCA; information of certain interest was survival, localization, initiation of bystander CPR and actions from EMS personnel.

Identification of subgroups

Within this diverse entity of OHCA's further investigation of subgroups are required. Through advanced text searches using a bag-of-words model within the prehospital medical record, cases of interest among the predefined subgroups will be identified; thus, is text-string searches developed for every subgroup. These predefined subgroups will be defined as trauma, drowning, electrocution, drug overdose and asphyxia (external) according to the Utstein template. The identified cases will be coupled to the national registry after external manual validation.

Variables included

* Age: Age will be defined as the subject age at the time of the event.
* Sex: Sex will be stated as either male, female or undetermined derived from personal identification numbers. Gender will be characterized based on EMS-charts, in those cases without an identification number.
* Initial rhythm: The initial rhythm will be defined as the first rhythm observed by EMS personnel, and categorized as either shockable, non-shockable (asystole), non-shockable (other) or undetermined.
* Etiology of cardiac arrest: Presumed causes will be stated as either presumed cardiac, other medical cause, trauma, drug overdose, drowning, electrocution or asphyxia (external).
* Location of Incidence: Location will be characterized as either residential area, outdoors and nature, private home or other.
* Observation of occurrence: Cardiac arrests will be defined as either unwitnessed, bystander witnessed or EMS-witnessed.
* Cardio-pulmonary-resuscitation: CPR will include bystander-initiated CPR and EMS treatment with CPR.
* Defibrillation and use of automatic external defibrillators: Defibrillation will include defibrillation by bystanders and/or EMS personnel. Use of AED's includes using the device also in the case it did not deliver shocks.
* EMS-response time: This will be defined as the time between a dispatcher receiving the emergency call and the arrival of the first EMS-personnel.
* Hospitalization: Hospitalization will be considered as either; transported to hospital or declared dead by EMS-personnel.
* Return-of-spontaneous-circulation (ROSC): ROSC will be classified as the achievement of ROSC anytime between recognition of the event and termination (defined as either hospital admission or declaration of death by EMS-personnel).
* State at hospital admission: State of the case upon arrival at the hospital will be defined as either ROSC or ongoing CPR.
* Survival: Survival will be defined as ROSC at the time of hospital admission, additionally 30-day survival will be included, this derived from data from the National Patient Registry.
* Airway management: This includes the airway manoeuvres performed on each case. It is defined by listing the use of airway adjuncts such as nasopharyngeal airway, oropharyngeal airway as well as endo-tracheal intubation, supraglottic airway device and isolated bag-valve-mask ventilation.
* Use of Medication: This includes a dichotomous (yes/no) variable based upon the potential administration of medication (ie epinephrine) for each case.

Analysis and Data Presentation

All data will be pseudo-anonymized, and all analyses will be accomplished on an aggregated nationwide level. Data is collected using the STROBE (STrengthening the Reporting of OBservational studies in Epidemiology) statement. The objective of this project is to clarify etiology, descriptive data and prehospital interventions of different subgroups of OHCA's. Descriptive statistics includes the above-mentioned variables labelled with absolute numbers and percentages. Comparative analyses will be carried out using non-parametric testing to examine subgroups. Forward logistic regression analysis will be performed for multivariate analysis. Within this multivariate logistic regression analysis both known and unknown variables will be processed. Odds ratio for survival will be calculated stratified by etiology, localization, bystander and EMS-actions.

Risk Management Strategy and Ethical Considerations Since it is registry-based research, there is no patient contact and of such no harm possible or further ethical considerations of concern. GDPR will be followed according to danish law and the studies will be registered at the Danish Data Protection Agency, capital region of Denmark. According to Danish legislation, register-based research does not require ethical committee approval nor patient consent.

Perspectives

This project provides novel information regarding these subgroups of OHCA; The way of using artificial intelligence within text mining allows high quality use of data in order to strengthen the results. Thus, the descriptive statistics provides relevant data based on a reviewed, high-quality database. Furthermore, throughout analyses, a better understanding of the preceding circumstances, etiology and prehospital assessment might contribute to improve handling these types of arrests. This, eventually through use of campaigns, education and training targeted laypersons and healthcare personnel, respectly.

Publication The results are targeted for publication in an international peer reviewed journal. Signe Amalie Wolthers is primary investigator of this project and will be listed as first author. Participation as coauthors will be decided according to the Vancouver criteria or acknowledged for providing access to data. All Danish regional EMS regions will receive this manuscript prior to publication for eventual comments.

ELIGIBILITY:
OHCA from non-cardiac origin

Inclusion Criteria:

* OHCA from non-cardiac origin (trauma, asphyxia, electrocution, drowning, overdose)

Exclusion Criteria:

* OHCA from cardiac origin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study evaluates OHCA from non-cardiac origin in the general population of Denmark between 2016 to 2021
Sampling Method: Probability Sample
Enrollment: 31200 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Survival | The timeframe is at the time of hospital admission, therefore no specific time point (ie 24-hours, 1hour ect) can be stated
  Status at admission. Categorical variable, polytomous outcome. (declared dead on scene, ongoing cpr, ROSC but unconscious, ROSC and aware)
longterm survival | 30 day
  30-day survival

SECONDARY OUTCOMES:
ROSC at any time | The timeframe is from incident (at scene) to admission to hospital. As of such it is not meassured at any specific time or time point, however the timeframe does not exceed 6 hours
  Return Of Spontanous Circulation at any time from incident to admission to hospital. It is a categorical variable with a binary outcome (yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- Prehospital Center, Næstved, Denmark

REFERENCES:
- [Background] Cummins RO, Chamberlain DA, Abramson NS, Allen M, Baskett PJ, Becker L, Bossaert L, Delooz HH, Dick WF, Eisenberg MS, et al. Recommended guidelines for uniform reporting of data from out-of-hospital cardiac arrest: the Utstein Style. A statement for health professionals from a task force of the American Heart Association, the European Resuscitation Council, the Heart and Stroke Foundation of Canada, and the Australian Resuscitation Council. Circulation. 1991 Aug;84(2):960-75. doi: 10.1161/01.cir.84.2.960. No abstract available. PMID 1860248
- [Background] Lindskou TA, Mikkelsen S, Christensen EF, Hansen PA, Jorgensen G, Hendriksen OM, Kirkegaard H, Berlac PA, Sovso MB. The Danish prehospital emergency healthcare system and research possibilities. Scand J Trauma Resusc Emerg Med. 2019 Nov 4;27(1):100. doi: 10.1186/s13049-019-0676-5. PMID 31684982
- [Background] Claesson A, Djarv T, Nordberg P, Ringh M, Hollenberg J, Axelsson C, Ravn-Fischer A, Stromsoe A. Medical versus non medical etiology in out-of-hospital cardiac arrest-Changes in outcome in relation to the revised Utstein template. Resuscitation. 2017 Jan;110:48-55. doi: 10.1016/j.resuscitation.2016.10.019. Epub 2016 Nov 5. PMID 27826118
- [Background] Christensen DM, Rajan S, Kragholm K, Sondergaard KB, Hansen OM, Gerds TA, Torp-Pedersen C, Gislason GH, Lippert FK, Barcella CA. Bystander cardiopulmonary resuscitation and survival in patients with out-of-hospital cardiac arrest of non-cardiac origin. Resuscitation. 2019 Jul;140:98-105. doi: 10.1016/j.resuscitation.2019.05.014. Epub 2019 May 23. PMID 31129226
- [Background] Lott C, Truhlar A, Alfonzo A, Barelli A, Gonzalez-Salvado V, Hinkelbein J, Nolan JP, Paal P, Perkins GD, Thies KC, Yeung J, Zideman DA, Soar J; ERC Special Circumstances Writing Group Collaborators. European Resuscitation Council Guidelines 2021: Cardiac arrest in special circumstances. Resuscitation. 2021 Apr;161:152-219. doi: 10.1016/j.resuscitation.2021.02.011. Epub 2021 Mar 24. PMID 33773826
- [Background] Kleber C, Giesecke MT, Lindner T, Haas NP, Buschmann CT. Requirement for a structured algorithm in cardiac arrest following major trauma: epidemiology, management errors, and preventability of traumatic deaths in Berlin. Resuscitation. 2014 Mar;85(3):405-10. doi: 10.1016/j.resuscitation.2013.11.009. Epub 2013 Nov 25. PMID 24287328
- [Background] Hess EP, Campbell RL, White RD. Epidemiology, trends, and outcome of out-of-hospital cardiac arrest of non-cardiac origin. Resuscitation. 2007 Feb;72(2):200-6. doi: 10.1016/j.resuscitation.2006.06.040. Epub 2006 Nov 22. PMID 17118509